CLINICAL TRIAL: NCT05956821
Title: Phase I/II Trial of Repeat Dosing of Super-Selective Intraarterial Infusion of Erbitux (Cetuximab) and Avastin (Bevacizumab) for Treatment of Relapsed/Refractory Intracranial Glioma in Patients Under 22 Years of Age
Brief Title: Treatment of Relapsed/Refractory Intracranial Glioma in Patients Under 22 Years of Age
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Heather McCrea, MD, Assistant Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20230032
Record Dates: First submitted 2023-07-14; First posted 2023-07-21 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma Multiforme; Anaplastic Astrocytoma; Fibrillary Astrocytomas; Oligodendroglioma; Diffuse Intrinsic Brainstem Glioma; Diffuse Intrinsic Pontine Glioma; DIPG Brain Tumor; H3 K27M
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Oligodendroglioma; Diffuse Intrinsic Pontine Glioma | interventions — Bevacizumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SIACI of cetuximab and bevacizumab (Experimental): Participants in this group will receive Cetuximab and Bevacizumab infusion into an artery each month for up to approximately one year.
  Interventions: Drug: SIACI of cetuximab and bevacizumab

INTERVENTIONS:
Drug: SIACI of cetuximab and bevacizumab — Subjects will receive monthly dosing of bevacizumab (15 mg/kg) and cetuximab (200mg/m2)
  Other Names: erbitux; avastin

SUMMARY:
This study assesses the safety and efficacy of repeat monthly dosing of super-selective intra-arterial cerebral infusion (SIACI) of cetuximab and bevacizumab in patients < 22 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Documented histologic diagnosis of relapsed or refractory glioblastoma multiforme (GBM), anaplastic astrocytoma (AA), fibrillary astrocytomas (FA), pilomyxoid astrocytoma (PXA), oligodendroglioma, or anaplastic mixed oligoastrocytoma (AOA), or radiologically diagnosed diffuse intrinsic brainstem glioma (DIPG)
* Must have at least one confirmed and evaluable tumor site
* Must have a Karnofsky or Lansky performance status ≥60%.
* No chemotherapy for three weeks prior to treatment
* Patients must have adequate hematologic reserve with absolute neutrophils≥1000/mm3 and platelets ≥100,000/ mm3
* Pre-enrollment chemistry parameters must show: bilirubin<1.5x the institutional upper limit of normal (IUNL); Aspartate Aminotransferase( AST) or Alanine transaminase (ALT)<2.5x IUNL and creatinine<1.5x IUNL
* Pre-enrollment coagulation parameters (PT and PTT) must be ≤1.5x the IUNL
* Growth factor(s): Must not have received within 1 week of entry onto this study
* Steroids: Systemic corticosteroid therapy is permissible in patients with Central Nervous System (CNS) tumors for treatment of increased intracranial pressure or symptomatic tumor edema. Patients with CNS tumors who are receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to study entry.
* Patients of reproductive age must agree to use a medically effective method of contraception during and for a period of three months after the treatment period. A pregnancy test will be performed on each premenopausal female of childbearing potential immediately prior to entry into the research study
* Patients or their parents/guardians must be able to understand and give written informed consent. Informed consent must be obtained at the time of patient screening
* Because of known concerns with Avastin and wound healing, craniotomy patients are eligible for the treatment if they have had a craniotomy greater than two weeks prior to Intra-Arterial (IA) therapy. Craniotomy or major procedure after SIACI Avastin therapy should wait 4 weeks. Minor surgeries may be performed after two weeks

Exclusion Criteria:

* Females who are pregnant or lactating
* Females of childbearing potential and fertile men will be informed as to the potential risk of procreation while participating in this research trial and will be advised that they must use effective contraception during and for a period of three months after the treatment period. If they do not agree, they will be ineligible for the study
* Patients with significant concurrent medical or psychiatric conditions that would place them at increased risk or affect their ability to receive or comply with treatment or post-treatment clinical monitoring

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2029-10-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Treatment Related Adverse Events | 1 month post injection
  The number of treatment-related adverse events will be assessed and graded according to the NCI Common Toxicity Criteria, version 5.0.
Composite Overall Response Rate (CORR) | 6 months
  The overall response proportion along with a 95% confidence interval will be estimated via binomial proportions. We will define "evaluable" patients as patients who met eligibility requirements and have initiated therapy.
Progression-free survival (PFS) | 1 year
  PFS will be measured from the date of the first dose of SIACI Cetuximab/Avastin to the date of progression.
Overall Survival (OS) | 1 year
  OS will be measured from the date of diagnosis to the date of death

CONTACTS AND LOCATIONS:
Overall Officials: Heather McCrea, MD, Principal Investigator — University of Miami
Locations (1):
- Jackson Memorial Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCrea HJ, Ivanidze J, O'Connor A, Hersh EH, Boockvar JA, Gobin YP, Knopman J, Greenfield JP. Intraarterial delivery of bevacizumab and cetuximab utilizing blood-brain barrier disruption in children with high-grade glioma and diffuse intrinsic pontine glioma: results of a phase I trial. J Neurosurg Pediatr. 2021 Aug 6;28(4):371-379. doi: 10.3171/2021.3.PEDS20738. Print 2021 Oct 1. PMID 34359048